CLINICAL TRIAL: NCT02714621
Title: Magnetic Resonance Guided High Intensity Focused Ultrasound (MRgHIFU): A Feasibility Study for Treating Recurrent Gynaecological Malignancies
Brief Title: MR-HIFU for Recurrent Gynaecological Cancer
Acronym: HIFU-Gynae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15/WM/0470 CCR4360
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Cervical Cancer; Endometrial Cancer; Uterine Cancer; Ovarian Cancer; Vaginal Cancer; Vulvar Cancer
Keywords: Magnetic Resonance Imaging (MRI); High Intensity Focused Ultrasound (HIFU); Focused Ultrasound Surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

ARMS (2):
- Feasibility of MR-HIFU for painful gynaecological metastases (No Intervention): Investigating whether it would be possible to use the MRgHIFU system to treat recurrent gynaecological cancers.
- Treatment using MR-HIFU of painful gynaecological metastases (Experimental): Testing whether MRgHIFU could be an effective treatment for the symptoms of recurrent gynaecological cancers (pain and bleeding)
  Interventions: Device: Magnetic Resonance Image-guided High Intensity Focused Ultrasound (MR-HIFU)

INTERVENTIONS:
Device: Magnetic Resonance Image-guided High Intensity Focused Ultrasound (MR-HIFU)
  Arms: Treatment using MR-HIFU of painful gynaecological metastases

SUMMARY:
The primary objective of this pilot study is to determine whether or not it is feasible to use MRgHIFU to treat symptomatic (pain, bleeding) recurrent pelvic malignancy with an acceptable safety profile when conventional treatment options are not available. The ultimate goal is to be able not only to offer a viable method of symptom palliation in patients with recurrent pelvic tumours and improve their quality of life; but also to control tumour growth and extend life in a group of relatively young patients with isolated local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent pelvic gynaecological malignancy (cervix and endometrial cancer).
* Recurrent lesion is painful (NRS>4) and not suitable for alternative treatments
* Intended target volume accessible for MRgHIFU treatment
* Intended target volume visible on noncontrast MR imaging
* Distance between target and skin ≥1cm

Exclusion Criteria:

* MRI contraindicated (e.g. by incompatible metal implants or claustrophobia)
* Pregnancy
* Sedation contraindicated
* MRI contrast agent contraindicated
* Scar, internal or external fixation device along the beam path or at the target

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in pain, measured using a patient diary | 7 days post-treatment, follow up at 90 days

SECONDARY OUTCOMES:
Changes in bleeding, measured using a questionnaire | 7 days post-treatment, follow up at 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Imseeh G, Giles SL, Taylor A, Brown MRD, Rivens I, Gordon-Williams R, Ter Haar G, deSouza NM. Feasibility of palliating recurrent gynecological tumors with MRGHIFU: comparison of symptom, quality-of-life, and imaging response in intra and extra-pelvic disease. Int J Hyperthermia. 2021;38(1):623-632. doi: 10.1080/02656736.2021.1904154. PMID 33882792